CLINICAL TRIAL: NCT02002065
Title: The Phase IV, Open-labelled, Follow-up Study to Evaluate the Five-year Immune Persistence of One Injection of Inactivated or Attenuated Alive Hepatitis A Vaccine in Healthy Chinese Children
Brief Title: The Fifth-year Follow-up Study for the Phase IV Clinical Trial of Hepatitis A Vaccine in Healthy Children
Status: Completed | Type: Observational
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-HA-4013 version 2.0
Record Dates: First submitted 2013-11-28; First posted 2013-12-05 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-04

CONDITIONS: Hepatitis A
Keywords: hepatitis A; inactivated hepatitis A vaccine; attenuated alive hepatitis A vaccine; immune persistence
MeSH Terms: conditions — Hepatitis A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples were taken from subjects.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Inactivated HAV vaccine: Inactivated vaccine: 0.5 ml per dose containing 250 u antigen, one dose
  Interventions: Biological: Inactivated HAV vaccine
- Attenuated alive HAV vaccine: Attenuated alive vaccine: 1.0 ml per dose containing 6.50 lgCCID50 alive virus, one dose
  Interventions: Biological: Attenuated alive HAV vaccine

INTERVENTIONS:
Biological: Inactivated HAV vaccine — Inactivated vaccine: 0.5 ml per dose containing 250 u antigen, one dose
  Groups: Inactivated HAV vaccine
Biological: Attenuated alive HAV vaccine — Attenuated alive vaccine: 1.0 ml per dose containing 6.50 lgCCID50 alive virus, one dose
  Groups: Attenuated alive HAV vaccine

SUMMARY:
The purpose of this follow-up study is to evaluate the five-year immune persistence of one injection of inactivated and attenuated alive hepatitis A vaccine in healthy children.

DETAILED DESCRIPTION:
In the previous double-blind, randomized, phase IV clinical trial in 2008, 300 healthy Chinese children aged 18 to 35 months old were administered with one dose of inactivated and attenuated alive hepatitis A vaccine. Series of serum samples were taken for immunogenicity and immune persistence evaluation. Safety observations were performed after vaccination. This trial was also approved by Tianjin CDC Biomedical Ethics Committee in 2008.

This study is the fifth-year follow-up research for the previous clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* All subjects who received inactivated or attenuated alive HAV vaccine in the previous trial

Exclusion Criteria:

* Subjects who refused to continue in the follow-up study

Ages: 18 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy Chinese children aged 18 to 35 months old
Sampling Method: Non-Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2008-10; Primary Completion 2013-11 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The geometric mean concentration (GMC) of anti-hepatitis A virus (HAV) antibodies in serum 60 months after vaccination | 60 months after vaccination
  to evaluate the immune persistence of anti-HAV antibodies in serum

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Lun Zhang, Principal Investigator — Tianjin Center for Diseases Control and Prevention
Locations (1):
- Tianjin center for disease prevention and control, Tianjin, China

REFERENCES:
- [Derived] Zhang Z, Zhu X, Hu Y, Liang M, Sun J, Song Y, Yang Q, Ji H, Zeng G, Song L, Chen J. Five-year antibody persistence in children after one dose of inactivated or live attenuated hepatitis A vaccine. Hum Vaccin Immunother. 2017 Jun 3;13(6):1-6. doi: 10.1080/21645515.2016.1278329. Epub 2017 Feb 14. PMID 28319454